CLINICAL TRIAL: NCT04838015
Title: Retrospective Study on Registry Data to Evaluate the Impact of Ocrelizumab Used in Routine Care in Patients With RRMS
Acronym: SEP-RR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8037
Record Dates: First submitted 2021-02-26; First posted 2021-04-08 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: MS-RR; Ocrelizumab; Switch
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple Sclerosis (MS) is a chronic, autoimmune, neurodegenerative disease; clinical events are mainly attributed to myelin destruction and inflammatory of the central nervous system.

The diagnosis resides in clinical and radiological criteria according to 2017 McDonald criteria.

Once the diagnosis of MS has been made, treatment should be initiated promptly, in order to delay the onset of severe disability in the long-term, even more ocrelizumab are a treatment of high efficacy.

Ocrelizumab is used as a first-line or second-line treatment in Relapsing Remitting MS (RRMS) It is an anti-CD20 monoclonal antibody that provides rapid depletion of circulating CD20+ B lymphocytes by complement-dependent cytotoxicity and antibody-dependent cellular cytotoxicity.

The main objective is the retrospective evaluation of the impact of ocrelizumab on the outcome of MS.

The secondary objective is the search of predictive factors of response to treatment.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Suffering from relapsing-remitting MS (RRMS)
* Supported in a neurology department at Strasbourg or Nancy University Hospital between 10/01/2018 and 11/31/2020.
* Treated with ocrelizumab 600mg every 6 months during the period from 01/10/2018 to 01/05/2020.
* Have had an M0, M3 / M6 and M12 MRI after initiation of treatment.
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Primary progressive multiple sclerosis (MS-PP), secondarily progressive (MS-SP)
* Subject not meeting all the inclusion criteria
* Impossibility of providing the subject with enlightened information (difficulties in understanding the subject, etc.)
* Subjects under safeguard of justice
* Subject under guardianship or guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject Suffering from relapsing-remitting MS
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-11-13 (Estimated); Study Completion 2021-11-13 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the impact of ocrelizumab used in patients with multiple sclerosis | Files analysed retrospectively from October 01, 2018 to November 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Hautepierre Clinical Investigation Center - Strasbourg University Hospitals, Strasbourg, France